CLINICAL TRIAL: NCT02840604
Title: What Benefit of a Full Analysis of Exome? Routine Care Study in Patients With Solid Tumors
Acronym: EXOMA
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: EXOMA
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient with all types of solid malignant tumors not treatable: In the treatment or assessment of metastatic solid tumor malignancies not curable it can be offered to patients to establish the profile of their tumor by next generation sequencing (NGS). This technique permits the sequencing of millions of fragments in parallel in a short time and allows to identify rapidly somatic or constitutional mutations known or yet unknown. The establishment of the genetic profile of the tumor coupled to the available clinical data can help clinicians to predict patient outcome in terms of survival or progression to disease, but may also provide key clues to adapt the management and patient treatment.

SUMMARY:
The management of cancers and their therapeutic guidance was until shortly mostly based on histopathological considerations of the tumor. the development of targeted therapies is a turning point and keeps increase. These molecules target a specific molecular defect in the tumor making it more effective and more specific treatment. But these treatments are only effective if the tumor has a specific molecular abnormality that is characterized and known.

These therapeutic progresses have been made possible through the decoding of the human genome and the molecular defects occurring during the carcinogenesis process. Now, dozens of therapies targeting a specific molecular abnormality are available in the therapeutic arsenal and dozens more are under development in clinical trials Phase 1 to 3.

In recent years, the democratization of next generation sequencing has opened a new era in cancer research but also for molecular diagnostics. Indeed, the enormous sequencing capabilities offered by high-throughput sequencing technologies allow analysis in a limited time the entire coding sequence of the genome (exome), or even the entire genome of a tumor (whole genome sequencing). Thus, the evolution and the development of broadband and associated bioinformatics tools for genomics techniques now make it possible to establish the genetic profile of a tumor. Targeted diagnosis of molecular abnormalities and allows to propose and specifically targeted direct therapeutic identified genetic alterations and supposedly responsible for tumor development. An analysis of tumor exome by next-generation sequencing (NGS) and provides information on genetic modifications of these tumors.

This study did not aim to evaluate a therapeutic strategy or treatment. The objective of this study is to evaluate the clinical benefit of an analysis of exome performed in current practice at the Centre Georges-François Leclerc from Dijon. The analysis will be performed by quantifying the number of patients undergoing therapeutic proposal based on the results of the analysis of the profile of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* histological and cytological diagnosis of solid evidence of malignancy metastatic or locally advanced non-curable and non-curable
* Disease for which a treatment under the national standards do not exist or will not exist if it escapes the current treatment
* Availability of equipment or new tumor biopsy / puncture a feasible accessed injury (biopsiable disease), only if it is deemed necessary in the treatment by the investigator.
* Patient affiliated with a social security scheme
* Patient non opposition

Exclusion Criteria:

* No tumor material available for the establishment of the tumor profile.
* Patient refusal
* Psychiatric illness and / or patient condition compromising the understanding of the information or the conduct of the study
* Patient under guardianship or subject to major people protection regime

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with all types of solid malignant tumors not treatable metastatic
Sampling Method: Probability Sample
Enrollment: 795 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of exome analysis for patient with a malignant solid tumors | 1 month
  Feasibility assess by whether or not the patient will have targeted therapeutic

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, Pr, Study Director — Centre Georges François Leclerc
Locations (1):
- CGFL, Dijon, France

REFERENCES:
- [Derived] Ratovomanana T, Cohen R, Svrcek M, Renaud F, Cervera P, Siret A, Letourneur Q, Buhard O, Bourgoin P, Guillerm E, Dorard C, Nicolle R, Ayadi M, Touat M, Bielle F, Sanson M, Le Rouzic P, Buisine MP, Piessen G, Collura A, Flejou JF, de Reynies A, Coulet F, Ghiringhelli F, Andre T, Jonchere V, Duval A. Performance of Next-Generation Sequencing for the Detection of Microsatellite Instability in Colorectal Cancer With Deficient DNA Mismatch Repair. Gastroenterology. 2021 Sep;161(3):814-826.e7. doi: 10.1053/j.gastro.2021.05.007. Epub 2021 May 13. PMID 33992635